CLINICAL TRIAL: NCT02698319
Title: The Copenhagen Triage Algorithm
Acronym: CTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Rasmus Bo Hasselbalch, Medical student, Herlev Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HerlevH02
Record Dates: First submitted 2016-02-24; First posted 2016-03-03 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Triage
Keywords: Triage; Systematic Triage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Triage (No Intervention): Conventional triage using Danish Emergency Process Triage (DEPT).
- Copenhagen Triage Algorithm (Experimental): The Copenhagen Triage Algorithm is used as triage form in the ED. The Copenhagen Triage Algorithm consists of a few vital parameters and a clinical assessment from the ED nurse.
  Interventions: Behavioral: Copenhagen Triage Algorithm

INTERVENTIONS:
Behavioral: Copenhagen Triage Algorithm — The Copenhagen Triage Algorithm is a new triage method for faster triage in the ED
  Arms: Copenhagen Triage Algorithm

SUMMARY:
Crowding in the emergency department (ED) is a well documented problem putting patients at risk of adverse outcomes. To combat this, most ED's use some form of triage. In the last two decades systematic triage or process triage has become the norm in most countries but this approach is supported by limited evidence. Our aim is to develop a faster triage model of only a few vital parameters, based on a data from a large cohort of unselected ED patients and evaluate if such a model combined with a clinical assessment by the ED nurse is inferior to existing triage models in a prospective cluster-randomized trial

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting acutely to the Acute ward/Emergency department in two hospitals in the Capital of Denmark

Exclusion Criteria:

* Patients presenting in Pediatric, Gynecological or Obstetric units

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50000 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 30 days
  Time frame starts at the beginning of the index admission, defined as first admission in the study period. Patients will be followed using central registers.

SECONDARY OUTCOMES:
Number of patients with an admission to the intensive care unit | 30 days
Length of stay during admission | 30 days
Waiting time for treatment | 8 hours
  Waiting time from first presenting at ED to first treatment startet
Number of readmissions | 30 and 90 days
  Patients will be followed using central registers. All new admissions within 91 days of the same patient is defined as readmissions.
All cause mortality | 48 hours
All cause mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Kasper Iversen, MD, DMSci, Principal Investigator — kasper.karmark.iversen@regionh.dk
Locations (2):
- Denmark (2):
  - Herlev Hospital, Herlev, Capital Region
  - Bispebjerg Hospital, København NV, Capital Region

REFERENCES:
- [Derived] Andrea MK, Pries-Heje M, Hasselbalch RB, Schultz M, Ravn L, Lind M, Christensen AH, Dalsgaard M, Iversen K. Causes of death among non-urgent patients in the emergency department who die within 30 days. Dan Med J. 2023 Sep 25;70(10):A01230037. PMID 37897388
- [Derived] Hasselbalch RB, Pries-Heje M, Schultz M, Plesner LL, Ravn L, Lind M, Greibe R, Jensen BN, Hoi-Hansen T, Carlson N, Torp-Pedersen C, Rasmussen LS, Iversen K. The Copenhagen Triage Algorithm is non-inferior to a traditional triage algorithm: A cluster-randomized study. PLoS One. 2019 Feb 4;14(2):e0211769. doi: 10.1371/journal.pone.0211769. eCollection 2019. PMID 30716123
- [Derived] Hasselbalch RB, Plesner LL, Pries-Heje M, Ravn L, Lind M, Greibe R, Jensen BN, Rasmussen LS, Iversen K. The Copenhagen Triage Algorithm: a randomized controlled trial. Scand J Trauma Resusc Emerg Med. 2016 Oct 10;24(1):123. doi: 10.1186/s13049-016-0312-6. PMID 27724978